CLINICAL TRIAL: NCT03310372
Title: Phase II Clinical Trial of Concomitant Association of Ultrafractionated Brain Irradiation - Temozolomide in Inoperable Primary Glioblastoma Multiforme
Brief Title: Concomitant Association of Ultrafractionated Brain Irradiation - Temozolomide in Inoperable Primary Glioblastoma Multiforme
Acronym: TEMOFRAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-004968-41
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrafractionated brain irradiation - temozolomide (Experimental)
  Interventions: Radiation: Ultrafractionated brain irradiation; Drug: Temozolomide

INTERVENTIONS:
Radiation: Ultrafractionated brain irradiation — 0.75 Gy a day, 5 times a week, for 6 weeks (total dose: 67.5 Gy)
Drug: Temozolomide — 75 mg/m2/day, 7 times a week, for 6 weeks (total 42 days)
  Other Names: Temodal

SUMMARY:
The main purpose of this study is the evaluation of concomitant association of ultrafractionated irradiation and Temodal® in patients with inoperable primary glioblastoma multiforme; study of tolerance and objective response rate.

The secondary purposes of this study are the evaluation of progression free survival, global survival and tolerance through toxicity study. The therapeutic response according to methylation or not of MGMT is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* giving their informed consent
* having a supratentorial malignant glioma, either grade 4 of St. Anne/Mayo grading, or glioblastoma multiforme according to WHO classification
* having an inoperable brain tumor (diagnosed by stereotactic biopsy)
* having a general status, evaluated by Karnofsky scale, >60
* having a life expectancy >3 months
* not having previously had a brain irradiation and/or adjuvant or neo-adjuvant chemotherapy
* potentially having another cancer, if histology and clinical history are available for comparison
* being able to take oral tablets
* no HIV disease
* satisfactory hematology, hepatic and renal functions: polymorphonuclear neutrophils >1500/mm3, platelets >100000/mm3, Hb >8g/dl, creatinemia ≤1.5 times upper normal value, total bilirubin <1.5 times upper normal value, ASAT and ALAT <3 times upper normal value
* for women of childbearing potential, a contraception is given

Exclusion Criteria:

* having an under tentorial malignant glioma (brain stem and/or cerebellum), grade 4 of St. Anne/Mayo grading
* having a Karnofsky score <60
* having a life expectancy <3 months
* having had a brain irradiation or an adjuvant or neoadjuvant chemotherapy
* refusing any additional therapy
* having a non-malignant but serious systemic disease or uncontrolled active infection
* having a severe psychiatric disorder
* not having signed the informed consent
* pregnant or breastfeeding woman

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-02-13 (Actual); Primary Completion 2012-06-26 (Actual); Study Completion 2012-06-26 (Actual)

PRIMARY OUTCOMES:
complete response | through study completion, 2 years
  defined as total regression of tumor area contrast in MRI, with stability or amelioration of neurological status of patient without corticoids
partial response | through study completion, 2 years
  defined by at least 50% diminution of tumor size, evaluated by the product of 2 perpendicular diameters measured by MRI, with stability or amelioration of neurological status of patient receiving stable or reduced corticoid doses
stabilization | through study completion, 2 years
  corresponding to at least 50% diminution of tumor size in MRI, with stability of neurological status of patient receiving steady corticoid doses
progression | through study completion, 2 years
  defined by increase of at least 25% of tumor size and/or a second brain localization in MRI, with degradation of neurological status of patient

SECONDARY OUTCOMES:
global survival | through study completion, 2 years
treatment tolerance | through study completion, 2 years
  evaluated by general, neurological and hematological status, according to National Cancer Institute-Common toxicity criteria (NCI-CTC)
survival without tumor recurrence | through study completion, 2 years
  tumor recurrence detected with radiology examination
life quality | through study completion, 2 years
  evaluated with European Organization for Research and Treatment of Cancer (EORTC) core quality of life questionnaire (QLQ - C30)

IPD SHARING:
Plan to Share IPD: No